CLINICAL TRIAL: NCT04715594
Title: A Whole Population-based Study on COreaN NationwidE Claims daTa on Drug-Eluting Stent (CONNECT DES) Registry
Brief Title: CONNECT DES Registrty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Myeong-Ki Hong, Professor, Yonsei University
Other Study IDs: 4-2019-0596
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Stent Thrombosis; Coronary Artery Disease; Stent Stenosis; Myocardial Infarction; Ischemic Heart Disease
Keywords: coronary artery disease; drug-eluting stents; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CONNECT DES Registrty
  Interventions: Device: 1st-generation drug-eluting stent; Device: 2nd-generation drug-eluting stents

INTERVENTIONS:
Device: 1st-generation drug-eluting stent — Implantation of 1st-generation drug-eluting stent
Device: 2nd-generation drug-eluting stents — Implantation of 2nd-generation drug-eluting stent

SUMMARY:
To date, drug-eluting stents (DES) have become the standard of care in daily practice for the treatment of ischemic heart disease, by overcoming the risk of in-stent restenosis, a major issue raised in the bare-mare stents era. The application of potent anti-proliferative drugs and polymer structures that ensures sustained released of the drugs markedly reduced the neointimal hyperplasia, leading to much improved clinical outcomes compared with bare-metal stents. However, although first-generation sirolimus-eluting stents and paclitaxel-eluting stents significantly reduced the risk of in-stent restenosis and target-vessel revascularization, an augmented risk for very late stent thrombosis and fatal clinical events emerged as a new issue to be solved. Second- and newer- generation DESs adopted innovative stent platforms, novel stent materials, anti-proliferative drugs, and biocompatible polymers (including both durable and bioresorbable). Nowadays, numerous types of DESs (over 20 types) are available in clinical practice as well as bare-metal stents. However, little is known about the clinical outcome according to type of DESs in real-word practice. Given that many of recent randomized clinical trials (RCTs) demonstrate the 'non-inferiority' of brand-new DESs over older DESs in limited period time (usually for 1-year) in a selected patients eligible for RCTs, the real-world clinical outcomes according to type of DES implanted are still unveiled. Although, the question about the differential impact of generation of DES, type of biocompatible polymers (bioresorbable versus durable), thickness of stent struts and type of eluted anti-proliferative drugs are very important in clinical aspect of view, but there is little study conducted on all patients who are actually confronted in daily clinical practice.

Korea operates national insurance system that covers most of the Koreans (97.1%) that are strictly monitored by National Health Insurance Service (NHIS). Of note, the claims database of NHIS of Korea contains all information including the demographic characters of patietns, diagnosis codes (ICD-9 and ICD-10), type of procedures or surgeries and the medical devices utilized, death certificates that contains type of death, and the drugs prescribe in outpatient clinic and hospitals in a individual pill level, that enables monitoring for the drug compliance. This unique feature of NHIS database allows the investigators to gain access to the dose and duration of cardio-protective medications including anti-platelet agents, lipid-lowering agents, anti-hypertensive agents, glucose-lowering agents, nitrate donors, vasodilators, and others. Given the benefits of NHIS database of Korea, we would like to establish a whole-population registry, named as COreaN NationwidE Claims daTa on Drug-Eluting Stent Registry (CONNECT DES Registry). A comprehensive analysis of this data is expected to shed new light on the impact of type of DESs and drug use in real-world practice that could be fully revealed through RCTs.

DETAILED DESCRIPTION:
According to stringent policy of NHIS database to protect personal information, information regarding type of DES including the thickness of strut, eluted drugs, type of polymer, generation of the DES will be provided after sufficient encryption. Likewise, all information regarding drug prescription, including the total number of pills prescribed during the period, patients' compliance and dosage of drugs will be provided after sufficient encryption. After decrypting the information provided to establish a database suitable for analysis, all eligible patients will be divided into two or more groups according to the type of DES or drug use pattern after DES implantation, which include:

1. 1st-generation vs. 2nd-generation DES
2. Durable polymer vs. bioresorbable polymer 2nd-generaion DES
3. Ultra-thin strut vs. Conventional strut vs. Thick-strut DES
4. According to the type of eluted drugs
5. DAPT duration after DES implantation
6. Type of anti-platelet therapy after cessation of DAPT
7. Intensity of statin therapy after DES implantation
8. According to use of nitrate donor or vasodilator after DES implantation
9. Use of anti-hypertensive agents after DES implantation
10. Use of glucose-lowering agents in diabetic subset of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients who were over 20 years old at the implantation of DES and treated with DES between 1-January-2005 and 31-December-2016

Exclusion Criteria:

* Patients who died within 1 week after DES implantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 350,000 patients with DES implantation between 2005 and 2016 would be incorporated in the analyses from National Health Insurance Service (NHIS) database
Sampling Method: Non-Probability Sample
Enrollment: 350000 (Estimated)
Dates: Start 2019-08-11 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5 years
  Death from any cause

SECONDARY OUTCOMES:
Cardiovascular mortality | 5 years
  Confirmed by death certificate with cardiovascular related diagnosis
Myocardial infarction | 5 years
Cardiovascular mortality or myocardial infarction | 5 years
  A composite of cardiovascular mortality and myocardial infarction
Ischemic Stroke | 5 years
Hemorrhagic stroke | 5 years
Any Stroke | 5 years
  A composite of ischemic stroke and hemorrhagic stroke
Gastrointestinal bleeding | 5 years
Any bleeding | 5 years
  Any bleeding
Major bleeding | 5 years
  Any bleeding that requires transfusion ≥2 units of red-blood cells, hospitalizaiton, procedure, surgery, or leading to disability or death
Net adverse clinical events (NACE) | 5 years
  A composite of all-cause mortality, recurrent MI, revascularization, ischemic stroke, and major bleeding
Major adverse cardiac events (MACE) | 5 years
  A composite of all-cause mortality, recurrent MI, and revascularization
Major adverse cardiac and cerebrovascular events (MACCE) | 5 years
  A composite of all-cause mortality, recurrent MI, revascularization, and ischemic stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Myeong-Ki, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Impossible to share the data due to goverment policy

REFERENCES:
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Background] Camenzind E, Steg PG, Wijns W. Stent thrombosis late after implantation of first-generation drug-eluting stents: a cause for concern. Circulation. 2007 Mar 20;115(11):1440-55; discussion 1455. doi: 10.1161/CIRCULATIONAHA.106.666800. Epub 2007 Mar 7. No abstract available. PMID 17344324
- [Background] Bangalore S, Toklu B, Patel N, Feit F, Stone GW. Newer-Generation Ultrathin Strut Drug-Eluting Stents Versus Older Second-Generation Thicker Strut Drug-Eluting Stents for Coronary Artery Disease. Circulation. 2018 Nov 13;138(20):2216-2226. doi: 10.1161/CIRCULATIONAHA.118.034456. PMID 29945934
- [Background] Kim D, Yang PS, Sung JH, Jang E, Yu HT, Kim TH, Uhm JS, Kim JY, Pak HN, Lee MH, Lip GYH, Joung B. Less dementia after catheter ablation for atrial fibrillation: a nationwide cohort study. Eur Heart J. 2020 Dec 14;41(47):4483-4493. doi: 10.1093/eurheartj/ehaa726. PMID 33022705
- [Derived] Lee SJ, Joo JH, Park S, Kim C, Choi DW, Lee YJ, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Nam CM, Hong MK. Combination therapy with moderate-intensity atorvastatin and ezetimibe vs. high-intensity atorvastatin monotherapy in patients treated with percutaneous coronary intervention in practice: assessing RACING generalizability. Eur Heart J Cardiovasc Pharmacother. 2025 Jan 11;10(8):676-685. doi: 10.1093/ehjcvp/pvad083. PMID 37951292
- [Derived] Lee SJ, Joo JH, Park S, Kim C, Choi DW, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Nam CM, Hong MK. Combination Lipid-Lowering Therapy in Patients Undergoing Percutaneous Coronary Intervention. J Am Coll Cardiol. 2023 Aug 1;82(5):401-410. doi: 10.1016/j.jacc.2023.05.042. PMID 37495276
- [Derived] Lee SJ, Choi DW, Kim C, Suh Y, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Park EC, Jang Y, Nam CM, Hong MK. Prolonged dual antiplatelet therapy after drug-eluting stent implantation in patients with diabetes mellitus: A nationwide retrospective cohort study. Front Cardiovasc Med. 2022 Aug 11;9:954704. doi: 10.3389/fcvm.2022.954704. eCollection 2022. PMID 36035946
- [Derived] Kim C, Choi DW, Lee SJ, Suh Y, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Park EC, Jang Y, Nam CM, Hong MK. Benefit and risk of prolonged dual antiplatelet therapy after drug-eluting stent implantation in patients with chronic kidney disease: A nationwide cohort study. Atherosclerosis. 2022 Jul;352:69-75. doi: 10.1016/j.atherosclerosis.2022.05.019. Epub 2022 Jun 8. PMID 35714431
- [Derived] Lee SJ, Choi DW, Kim C, Suh Y, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Park EC, Jang Y, Nam CM, Hong MK. Long-Term Beta-Blocker Therapy in Patients With Stable Coronary Artery Disease After Percutaneous Coronary Intervention. Front Cardiovasc Med. 2022 May 17;9:878003. doi: 10.3389/fcvm.2022.878003. eCollection 2022. PMID 35656394
- [Derived] Lee SJ, Choi DW, Suh Y, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Park EC, Jang Y, Nam CM, Hong MK. Long-Term Clinical Outcomes Between Biodegradable and Durable Polymer Drug-Eluting Stents: A Nationwide Cohort Study. Front Cardiovasc Med. 2022 Apr 29;9:873114. doi: 10.3389/fcvm.2022.873114. eCollection 2022. PMID 35571196